CLINICAL TRIAL: NCT04084860
Title: The Role of Brief Potent Glutamatergic Modulation in Addressing Problem Drinking: a Randomized, Controlled Trial
Brief Title: The Role of Brief Potent Glutamatergic Modulation in Addressing Problem Drinking
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7889; 5R01AA027509-02 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CI-581a + MET/MBRP (Experimental): Administration of CI-581a during weeks 1 and 6 at 0.71 mg/kg in the context of a 12 wk outpatient treatment (behavioral treatment combination of MET/MBRP will be provided)
  Interventions: Drug: CI-581a; Behavioral: MBRP; Behavioral: MET
- CI-581a + Medication Management (Experimental): Administration of CI-581a during weeks 1 and 6 at 0.71 mg/kg in the context of a 12 wk outpatient treatment ( no MET/MBRP sessions will be provided, only general check-ins and psychiatrist visits)
  Interventions: Drug: CI-581a
- CI-581b + MET/MBRP (Active Comparator): Administration of CI-581b during weeks 1 and 6 at 0.0125 mg/kg in the context of a 12 wk outpatient treatment (behavioral treatment combination of MET/MBRP will be provided)
  Interventions: Drug: CI-581b; Behavioral: MBRP; Behavioral: MET
- CI-581b + Medication Management (Active Comparator): Administration of CI-581b during weeks 1 and 6 at 0.0125 mg/kg in the context of a 12 wk outpatient treatment (no MET/MBRP sessions will be provided, only general check-ins and psychiatrist visits)
  Interventions: Drug: CI-581b

INTERVENTIONS:
Drug: CI-581a — CI-581a during weeks 1 and 6 at 0.71 mg/kg
  Arms: CI-581a + MET/MBRP; CI-581a + Medication Management
Drug: CI-581b — CI-581b during weeks 1 and 6 at 0.0125 mg/kg
  Arms: CI-581b + MET/MBRP; CI-581b + Medication Management
Behavioral: MBRP — MBRP will help with maintaining use reduction/abstinence.In this trial, 3 sessions will occur in the first 2 weeks following the second infusion (weeks 6 and 7), while one session a week will be administered in the latter 5 weeks (weeks 8 through 12).
  Other Names: Mindfulness Based Relapse Prevention (MBRP)
  Arms: CI-581a + MET/MBRP; CI-581b + MET/MBRP
Behavioral: MET — MET may help with goal setting and enhancing engagement with MBRP. In this trial, a standard 5-week MET platform will be provided to individuals randomized to receive behavioral treatment, with an additional session after each infusion (7 sessions total).
  Other Names: Motivational Enhancement Therapy (MET)
  Arms: CI-581a + MET/MBRP; CI-581b + MET/MBRP

SUMMARY:
The proposed project tests the efficacy of glutamate modulators in non-depressed individuals with alcohol use disorder (AUD); the primary hypothesis is that the glutamate modulator being tested reduces heavy drinking days compared to the active control. It also aims to investigate, using a 2 by 2 factorial (2x2) design, the hypothesis that the effects of the glutamate modulator are enhanced when combined with behavioral treatment.

DETAILED DESCRIPTION:
Alterations in glutamate neurotransmission are an important target of pharmacotherapy for alcohol use disorder. Our investigations with glutamate modulators in drug and alcohol dependent individuals suggest that they may exert unique therapeutic effects on dependence-related vulnerabilities and may also address problem drinking in alcohol dependent individuals. The proposed project will expand on our prior research by testing the efficacy of glutamate modulators in a larger population of non-depressed individuals with alcohol use disorder (AUD); it also aims to investigate, using a 2 by 2 factorial (2x2) design, the hypothesis that the effects of the glutamate modulator are enhanced when combined with behavioral treatment. It, therefore, has the potential to deepen our understanding of the therapeutic role of glutamate modulators in AUD treatment, as well as to provide further evidence for the efficacy of this novel pharmacotherapy strategy in addressing problem use

ELIGIBILITY:
Inclusion Criteria:

1. Active alcohol use disorder, with at least 4 heavy drinking day over the past 7 days (greater than 4 drinks a day for males, greater than 3 drinks for females). In the case of the use of other drugs, alcohol is designated as the primary drug
2. Physically healthy
3. No adverse reactions to study medications
4. 21-70 years of age
5. Capacity to consent and comply with study procedures, including sufficient proficiency in English
6. Seeking to reduce or stop alcohol use

Exclusion Criteria:

1. Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, or any psychotic illness, including substance-induced psychosis
2. Physiological dependence on another substance, such as opioids or benzodiazepines, excluding caffeine, nicotine, and cannabis
3. Delirium, Dementia, Amnesia, Cognitive Disorders, or Dissociative disorders
4. Current suicide risk or a history of suicide attempt within the past year
5. Inability to safely initiate 24 hours of abstinence from alcohol, as evidenced by CIWA greater than 10 during screening; history of severe withdrawal phenomena over the past 6 months (e.g., inpatient stabilization, withdrawal-related seizure); or self-reported inability to maintain abstinence for 24 hours.
6. Pregnant or interested in becoming pregnant during the study period
7. Any of the following cardiac conditions: clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia, or mitral valve prolapse
8. Unstable physical disorders which might make participation hazardous such as hypertension (>160/90), anemia, active hepatitis or other liver disease (transaminase levels < 2-3 X the upper limit of normal will be considered acceptable), epilepsy, or untreated diabetes. Participants reporting HIV+ status will be asked to provide information about their current treatment, including all medications. Participants who are on the antiretroviral ritonavir (Norvir) will be excluded due to the possibility that study medications in combination with this medication may increase the risk of drug-induced hepatitis.
9. Previous history of misuse or abuse of study medications, and a history of an adverse reaction/experience with prior exposure to study medications
10. Recent history of significant violance
11. On psychotropic or other medications whose effect could be disrupted by participation in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Daily occurrence of Heavy Drinking Days (HDD) | 12 weeks
  Defined as >4 drinks/day for men; >3 drinks for women. Comparing this outcome between groups that receive CI-581a versus CI-581b, as well as between CI-581a groups.

SECONDARY OUTCOMES:
Daily occurrence of drinking days | 12 weeks
  Comparing this outcome in between group that received CI-581a versus CI-581b, as well as between CI-581a groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — NYSPI/Columbia
Locations (1):
- NYSPI, New York, New York, United States